CLINICAL TRIAL: NCT00687245
Title: A Randomized, Open-Label Study to Evaluate the Pharmacokinetics of Single Oral Doses of Esomeprazole Magnesium in Pediatric Patients 1 to 11 Years-Old Inclusive With Endoscopically-Proven Gastroesophageal Reflux Disease (GERD)
Brief Title: Pharmacokinetic Study of Esomeprazole Magnesium in Patients 1 to 11 Years-Old With Endoscopically-Proven Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Tore Lind, MD, Medical Science Director Nexium and GI Established Brands, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: D9614C00007
Record Dates: First submitted 2008-05-28; First posted 2008-05-30 (Estimated); Last update posted 2008-06-11 (Estimated); Status verified 2008-06

CONDITIONS: Endoscopically-Proven GERD; Reflux
Keywords: children; reflux; GERD; pediatric
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): esomeprazole magnesium 5 mg, weight 8 kg to < 20kg
  Interventions: Drug: esomeprazole magnesium
- 2 (Experimental): esomeprazole magnesium 10 mg, weight 8 kg to < 20kg
  Interventions: Drug: esomeprazole magnesium
- 3 (Experimental): esomeprazole magnesium 10 mg, weight > 20 kg
  Interventions: Drug: esomeprazole magnesium
- 4 (Experimental): esomeprazole magnesium 20 mg, weight > 20 kg
  Interventions: Drug: esomeprazole magnesium

INTERVENTIONS:
Drug: esomeprazole magnesium — capsules, oral, qd, one day
  Other Names: Nexium

SUMMARY:
The purpose of this study is to determine the area under the plasma concentration-time curve (AUC) of esomeprazole after single oral doses of 5 mg, 10 mg or 20 mg esomeprazole in pediatric patients 1 to 11 years-old inclusive with endoscopically-proven GERD.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to take solid or bland food (eg, applesauce).
* Patients must weigh at least 8 kg and at the investigator's discretion be able to undergo extraction of an adequate volume of blood.
* The patient's weight for height percentile should be less than the 90th percentile and/or the BMI must be between the 5th and 85th percentile for age.
* Patients must be diagnosed with endoscopically-proven GERD

Exclusion Criteria:

* Use of any other investigational compound or participation in another clinical trial within 28 days prior to the screening visit.
* History or presence of gastrointestinal, hepatic or renal disease or other conditions that could interfere with absorption, distribution, metabolism or excretion of esomeprazole.
* Unstable diabetes mellitus or history of seizure disorder.
* Any acute or chronic illness or a medical history, which in the opinion of the investigator and/or sponsor, could compromise the patient's safety or successful participation in the study.

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2006-08; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) of esomeprazole after single oral doses of 5 mg, 10 mg and 20 mg esomeprazole in pediatric patients 1 to 11 years old inclusive with endoscopically-proven GERD. | Day 1

SECONDARY OUTCOMES:
The AUC(0-t), Cmax, tmax, and apparent volume of distribution during terminal phase (Vλz/F) of esomeprazole after single oral doses of 5 mg, 10 mg and 20 mg esomeprazole in pediatric patients 1 to 11 years-old inclusive with endoscopically-proven GERD. | Day 1
AUC, AUC(0-t), Cmax, tmax, t1/2λz of the 5-hydroxy and sulphone metabolites of esomeprazole after a single oral dose of 5 mg, 10 mg, and 20 mg esomeprazole in pediatric patients 1 to 11 years-old inclusive with endoscopically-proven GERD. | Day 1
Safety and tolerability after a single oral dose of esomeprazole in pediatric patients 1 to 11 years old inclusive with endoscopically- proven GERD. | Day 1, Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Marta Illueca, Study Director — AstraZeneca; Lynne Durborow, Study Chair — AstraZeneca

REFERENCES:
- [Derived] Earp JC, Mehrotra N, Peters KE, Fiorentino RP, Griebel D, Lee SC, Mulberg A, Rohss K, Sandstrom M, Taylor A, Tornoe CW, Wynn EL, Van der Walt JS, Garnett C. Esomeprazole FDA Approval in Children With GERD: Exposure-Matching and Exposure-Response. J Pediatr Gastroenterol Nutr. 2017 Sep;65(3):272-277. doi: 10.1097/MPG.0000000000001467. PMID 27875488